CLINICAL TRIAL: NCT04646408
Title: Determinants of Cardiovascular Disease, Kidney Disease and Diabetes in People of African Ancestry With HIV (CKD Study)
Brief Title: Determinants of Cardiovascular Disease, Kidney Disease and Diabetes
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: King's College Hospital NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: KingCKD
Record Dates: First submitted 2020-09-09; First posted 2020-11-30 (Actual); Last update posted 2020-11-30 (Actual); Status verified 2020-08

CONDITIONS: Cardiovascular Diseases; Diabetes Mellitus; Chronic Kidney Diseases
Keywords: chronic kidney disease; cardiovascular disease; HIV; syndemic; diabetes
MeSH Terms: conditions — Cardiovascular Diseases; Diabetes Mellitus; Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — * CKD: creatinine, albuminuria [ACR], proteinuria [PCR]
  * Diabetes: glucose and HbA1c
  * Metabolic: full lipid profile incl. HDL-cholesterol, triglycerides]
  * If no recent measures available: HIV RNA, Haemoglobin, Platelets, Liver enzymes [AST, ALT and GGT]
  * Inflammatory biomarkers: C-reactive protein (CRP)
  * Samples for future biomarkers e.g. C-peptide and inflammatory markers
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Participants with CKD: Recruitment is from a cohort of HIV positive individuals of African ancestry with Chronic Kidney Disease CKD defined as eGFR <60 mL/min/1.73m2, and/or albumin/creatinine ratio >30 mg/mmol or protein/creatinine ratio >50 mg/mmol Anticipated n=75
- Participants with diabetes: Recruitment is from a cohort of HIV positive individuals of African ancestry with diabetes. Diabetes is defined as being on diabetic medications or HbA1c >48 mmol/mol.
  Anticipated n=75
- Participants with ischaemic heart disease/stroke: Recruitment is from a cohort of HIV positive individuals of African ancestry with previous ischaemic heart disease or stroke Anticipated n=50
- No CKD/DM/CVD cohort: Recruitment is from a cohort of HIV positive individuals of African ancestry who do not have CKD, diabetes or prior ischaemic heart disease/stroke.
  Anticipated n=200

SUMMARY:
Cardiovascular disease (CVD), chronic kidney disease (CKD), diabetes mellitus (DM) and HIV infection are long-term conditions (LTC) with major health implications for people of African ancestry. These LTC often arise in the setting of an adverse demographic, social, biologic and genetic environment, although this remains poorly understood.

The investigators plan to conduct a comprehensive syndemic evaluation in individuals with and without CVD, CKD and DM in people of African ancestry with HIV to obtain novel insights into the development of LTC in this population. In addition, the investigators will conduct focus groups to explore the role of syndemic factors in the development of LTC and develop and pilot an educational programme to improve knowledge about LTC in the African/Caribbean community.

DETAILED DESCRIPTION:
Black African/Caribbean Communities in South London are disproportionally affected by long-term conditions (LTC), with a higher prevalence and an earlier onset (by about 13 years) (1). This population experiences high rates of hypertension, obesity, diabetes mellitus (DM), chronic kidney disease (CKD), cardiovascular disease (CVD) including stroke, social deprivation, poor housing, and mental health conditions such as anxiety and depression (1). HIV infection is also considerably more common in Black African/Caribbean Communities in South London than in the general UK population (2,3) and gives rise to stigma and discrimination, low self-esteem, dysfunctional relationships and loneliness (4).

The relationship between hypertension, obesity, metabolic syndrome, diabetes mellitus and CKD is well recognised. In this population, 'hypertensive nephropathy' is about 10-fold more common than in Caucasians, with earlier onset of end stage kidney disease (ESKD) (5). Although hypertensive nephropathy in people of African ancestry was previously attributed to resistant hypertension, exacerbated by poor engagement with health care services and suboptimal adherence to antihypertensive therapy, there is emerging evidence of strong genetic susceptibility to CKD as a result of prevalent mutations in the apolipoprotein L1 (APOL1), glutathione-S-transferase-μ1 (GSTM1) genes or sickle cell trait (SCT) (6-12). However, despite their strong associations with CKD, many individuals with these genetic variants do not develop kidney disease, suggesting that additional (i) biologic (e.g. coinfections, inflammation), (ii) environmental factors (e.g. obesity, diabetes), and (iii) socio-economic aspects, (e.g. inadequate health care access, stigma) may contribute to the development or progression of CKD although this has not been well studied.

There is growing recognition of the important role of social determinants of health (SDH) and its impact across a wide range of health indicators, settings, and populations (13,14). The World Health Organization (WHO) refers to SDH as conditions to which people are born, grow, work, live and age, linked to personal circumstances and systems (e.g. social, economic and political policies/heath care systems) that influences their daily lives (15-16). The new conceptual framework of syndemics provide an opportunity to study diseases and health conditions in populations that are deepened by the social, economic, environmental and political environment of a given population (17). The definition of a syndemic is 'the presence of two or more disease states (anchored around a core disease, in our case HIV) that adversely interact with each other, negatively affecting the mutual course of each disease trajectory, enhance vulnerability, and which are more harmful by experienced inequities' (18). This approach of a so-called 'syndemic lens' may be helpful in our study to identify the associations between genetic, biologic and social factors that contribute to the development of CKD and DM in people with hypertension, obesity, sub-clinical CKD and/or metabolic syndrome. This systemic approach can offer a new understanding of diseases that can improve public health and treat individual patients at the same time (19).

South London has a large (>200,000) population of African and Caribbean ancestry who are disproportionally affected by HIV and experience a higher burden of CKD, DM and other LTC, often with earlier onset compared to white populations. The investigators aim to study the demographic, clinical, social and genetic factors that associate with CKD, DM and multiple LTC in people with HIV. CKD and DM are key LTC that associate with hypertension, obesity and cardiovascular disease, resulting in or contribute to functional impairment, polypharmacy and impaired bio-psycho-social health outcomes.

The HIV clinics in South London provide a unique opportunity to access a diverse African and Caribbean population of working age in whom LTC can be studied. People with HIV from black African/Caribbean communities experience a high degree of social and economic deprivation, stigma, anxiety and depression which are considered important syndemic factors in the development of LTC. CKD and DM are common LTC, highly relevant to the black population, and relatively early events in the development of multiple and disabling LTC, thus identifying a population for targeted interventions that may reduce the rate of progression from a single to multiple LTC.

HIV infection, itself a LTC, can be effectively controlled with antiretroviral therapy, affording normal life expectancy and interrupting onward transmission. Routine care includes 6-12 monthly assessments for other LTCs, providing opportunities for recruitment of well characterised populations unselected for specific co-morbid conditions.

No studies to date in the UK have examined the contribution of biologic, clinical, social and genetic factors to the development of LTC in African/Caribbean populations with HIV to date. The team will generate detailed information on factors that associate with CKD, DM, CVD and multiple LTC as well as hypertension, sub-clinical CKD, obesity and insulin resistance, which often precede the development of CKD, DM and other LTC in this population. This study is likely to identify novel associations which can be confirmed and further explored in subsequent studies of HIV positive and general African/Caribbean populations. Stored biological samples will allow us to explore pathogenetic mechanisms in subsequent studies.

Key barriers to uptake of existing and novel interventions include low literacy levels, low perception of quality of life, lack of knowledge of LTCs, etc. The investigators will explore how best to overcome these barriers in focus groups and develop a culturally sensitive educational programme, aiming to reach individuals in communities that tend to poorly engage with health care and preventive programmes.

ELIGIBILITY:
Inclusion Criteria:

1. Having previously participated in the GEN-AFRICA study
2. Aged 18-60 years

Exclusion Criteria:

1. Not having participated in the GEN-AFRICA study
2. Aged >60 years

Ages: 18 Months to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Participants will be sampled from an existing cohort from the GEN AFRICA (Genetics Markers of Kidney Disease Progression in People of African Heritage Study). 75 participants with CKD, 75 participants with diabetes, 50 participants with a history of ischaemic heart (IHD)disease/stroke and 200 participants without CKD, diabetes, IHD/stroke will be recruited.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2022-09-01 (Estimated); Study Completion 2022-10-01 (Estimated)

PRIMARY OUTCOMES:
Obsity | 24months
  • To describe, in African/Caribbean adults with HIV, demographic, clinical, social, biologic, genetic factors associated with CVD, CKD, DM and multiple LTC and the major clinical risk factors for these:
  1. Obesity
Hypertension | 24months
  • To describe, in African/Caribbean adults with HIV, demographic, clinical, social, biologic, genetic factors associated with CVD, CKD, DM and multiple LTC and the major clinical risk factors for these: 2. Hypertension
CKD | 24months
  • To describe, in African/Caribbean adults with HIV, demographic, clinical, social, biologic, genetic factors associated with CVD, CKD, DM and multiple LTC and the major clinical risk factors for these: 3. CKD
Metabolic Syndrome | 24months
  • To describe, in African/Caribbean adults with HIV, demographic, clinical, social, biologic, genetic factors associated with CVD, CKD, DM and multiple LTC and the major clinical risk factors for these: 4. Metabolic syndrome
Syndemic aspects and qualitative assessment of contextual factors associated with long term health conditions | 24months
  • To explore more subtle variations of contextual factors and experiences about the role of syndemic aspects and provide further insights that may have been missed by the "itemised" quantitative approach in outcome 1. (using validated tools such as DISCUS, HADS, EQ-5D-5L)
Educational | 24months
  • To develop and pilot an educational programme on an existing App to improve knowledge about CKD, DM and CVD in the local African/Caribbean community.

CONTACTS AND LOCATIONS:
Locations (1):
- King's College London, London, Apartment G02, Cordage House, United Kingdom

REFERENCES:
- [Background] 1. GSTT Charity report: From one to many. Exploring people's progression to multiple longterm conditions in an urban environment. Guy's and St. Thomas' Charity, London, July 2018. p10. 2. Public Health England. HIV in the UK 2016 report.
- [Background] 2. Public Health England. HIV in the UK 2016 report. https://assets.publishing.service.gov.uk/government/uploads/system/uploads/attachment _data/file/602942/HIV_in_the_UK_report.pdf
- [Background] 3. Public Health England. Hepatitis B in London 2016 data. https://assets.publishing.service.gov.uk/government/uploads/system/uploads/attachment _data/file/801174/London_hepatitis_B_report_2016.pdf
- [Background] 4. Public Health England. Positive Voices: The National Survey of People Living with HIV. Findings from the 2017 Survey. https://assets.publishing.service.gov.uk/government/uploads/system/uploads/attachment_data/file/857922/PHE_positive_voices_report_2019.pdf
- [Background] Saran R, Li Y, Robinson B, Abbott KC, Agodoa LY, Ayanian J, Bragg-Gresham J, Balkrishnan R, Chen JL, Cope E, Eggers PW, Gillen D, Gipson D, Hailpern SM, Hall YN, He K, Herman W, Heung M, Hirth RA, Hutton D, Jacobsen SJ, Kalantar-Zadeh K, Kovesdy CP, Lu Y, Molnar MZ, Morgenstern H, Nallamothu B, Nguyen DV, O'Hare AM, Plattner B, Pisoni R, Port FK, Rao P, Rhee CM, Sakhuja A, Schaubel DE, Selewski DT, Shahinian V, Sim JJ, Song P, Streja E, Kurella Tamura M, Tentori F, White S, Woodside K, Hirth RA. US Renal Data System 2015 Annual Data Report: Epidemiology of Kidney Disease in the United States. Am J Kidney Dis. 2016 Mar;67(3 Suppl 1):Svii, S1-305. doi: 10.1053/j.ajkd.2015.12.014. No abstract available. PMID 26925525
- [Background] Kopp JB, Nelson GW, Sampath K, Johnson RC, Genovese G, An P, Friedman D, Briggs W, Dart R, Korbet S, Mokrzycki MH, Kimmel PL, Limou S, Ahuja TS, Berns JS, Fryc J, Simon EE, Smith MC, Trachtman H, Michel DM, Schelling JR, Vlahov D, Pollak M, Winkler CA. APOL1 genetic variants in focal segmental glomerulosclerosis and HIV-associated nephropathy. J Am Soc Nephrol. 2011 Nov;22(11):2129-37. doi: 10.1681/ASN.2011040388. Epub 2011 Oct 13. PMID 21997394
- [Background] Tin A, Scharpf R, Estrella MM, Yu B, Grove ML, Chang PP, Matsushita K, Kottgen A, Arking DE, Boerwinkle E, Le TH, Coresh J, Grams ME. The Loss of GSTM1 Associates with Kidney Failure and Heart Failure. J Am Soc Nephrol. 2017 Nov;28(11):3345-3352. doi: 10.1681/ASN.2017030228. Epub 2017 Jul 18. PMID 28720685
- [Background] Lipkowitz MS, Freedman BI, Langefeld CD, Comeau ME, Bowden DW, Kao WH, Astor BC, Bottinger EP, Iyengar SK, Klotman PE, Freedman RG, Zhang W, Parekh RS, Choi MJ, Nelson GW, Winkler CA, Kopp JB; SK Investigators. Apolipoprotein L1 gene variants associate with hypertension-attributed nephropathy and the rate of kidney function decline in African Americans. Kidney Int. 2013 Jan;83(1):114-20. doi: 10.1038/ki.2012.263. Epub 2012 Jul 25. PMID 22832513
- [Background] Genovese G, Friedman DJ, Ross MD, Lecordier L, Uzureau P, Freedman BI, Bowden DW, Langefeld CD, Oleksyk TK, Uscinski Knob AL, Bernhardy AJ, Hicks PJ, Nelson GW, Vanhollebeke B, Winkler CA, Kopp JB, Pays E, Pollak MR. Association of trypanolytic ApoL1 variants with kidney disease in African Americans. Science. 2010 Aug 13;329(5993):841-5. doi: 10.1126/science.1193032. Epub 2010 Jul 15. PMID 20647424
- [Background] Chang J, Ma JZ, Zeng Q, Cechova S, Gantz A, Nievergelt C, O'Connor D, Lipkowitz M, Le TH. Loss of GSTM1, a NRF2 target, is associated with accelerated progression of hypertensive kidney disease in the African American Study of Kidney Disease (AASK). Am J Physiol Renal Physiol. 2013 Feb 15;304(4):F348-55. doi: 10.1152/ajprenal.00568.2012. Epub 2012 Dec 5. PMID 23220723
- [Background] Naik RP, Derebail VK, Grams ME, Franceschini N, Auer PL, Peloso GM, Young BA, Lettre G, Peralta CA, Katz R, Hyacinth HI, Quarells RC, Grove ML, Bick AG, Fontanillas P, Rich SS, Smith JD, Boerwinkle E, Rosamond WD, Ito K, Lanzkron S, Coresh J, Correa A, Sarto GE, Key NS, Jacobs DR, Kathiresan S, Bibbins-Domingo K, Kshirsagar AV, Wilson JG, Reiner AP. Association of sickle cell trait with chronic kidney disease and albuminuria in African Americans. JAMA. 2014 Nov 26;312(20):2115-25. doi: 10.1001/jama.2014.15063. PMID 25393378
- [Background] Naik RP, Irvin MR, Judd S, Gutierrez OM, Zakai NA, Derebail VK, Peralta C, Lewis MR, Zhi D, Arnett D, McClellan W, Wilson JG, Reiner AP, Kopp JB, Winkler CA, Cushman M. Sickle Cell Trait and the Risk of ESRD in Blacks. J Am Soc Nephrol. 2017 Jul;28(7):2180-2187. doi: 10.1681/ASN.2016101086. Epub 2017 Mar 9. PMID 28280138
- [Background] Braveman P, Gottlieb L. The social determinants of health: it's time to consider the causes of the causes. Public Health Rep. 2014 Jan-Feb;129 Suppl 2(Suppl 2):19-31. doi: 10.1177/00333549141291S206. PMID 24385661
- [Background] Braveman P, Egerter S, Williams DR. The social determinants of health: coming of age. Annu Rev Public Health. 2011;32:381-98. doi: 10.1146/annurev-publhealth-031210-101218. PMID 21091195
- [Background] Social Determinants of Health. World Health Organization (WHO).
- [Background] Mendenhall E, Kohrt BA, Norris SA, Ndetei D, Prabhakaran D. Non-communicable disease syndemics: poverty, depression, and diabetes among low-income populations. Lancet. 2017 Mar 4;389(10072):951-963. doi: 10.1016/S0140-6736(17)30402-6. PMID 28271846
- [Background] The Lancet. Syndemics: health in context. Lancet. 2017 Mar 4;389(10072):881. doi: 10.1016/S0140-6736(17)30640-2. No abstract available. PMID 28271823
- [Background] Singer M, Bulled N, Ostrach B, Mendenhall E. Syndemics and the biosocial conception of health. Lancet. 2017 Mar 4;389(10072):941-950. doi: 10.1016/S0140-6736(17)30003-X. PMID 28271845
- [Background] Tsai AC, Mendenhall E, Trostle JA, Kawachi I. Co-occurring epidemics, syndemics, and population health. Lancet. 2017 Mar 4;389(10072):978-982. doi: 10.1016/S0140-6736(17)30403-8. No abstract available. PMID 28271848
- [Background] Barbour RS (2010) Focus groups Qualitative Health Research Practice. Sage, London, pp 327-352.
- [Background] Malterud K. Qualitative research: standards, challenges, and guidelines. Lancet. 2001 Aug 11;358(9280):483-8. doi: 10.1016/S0140-6736(01)05627-6. PMID 11513933
- [Background] Braun, V. and V. Clarke (2006). Using thematic analysis in psychology. Qualitative Research in Psychology, 3 (2), 77-101.
- [Background] Seale, C. (1999). Doing Qualitative Research: a Practical Handbook, D. Silverman, ed., Sage Publications, London, pp. 73-85, 119-138, and 154-172.
- [Background] Sousa D (2014). Validation in Qualitative Research: General Aspects and Specificities of the Descriptive Phenomenological Method, Qualitative Research in Psychology, 11:2, 211-227.